CLINICAL TRIAL: NCT06773260
Title: Assessment of Liver and Spleen Stiffness Measurement (LSM/SSM) Accuracy in Predicting the Presence of Oesophageal Varices Needing Treatment in Cirrhotic Patients With Advanced Hepatocellular Carcinoma (HCC) Who Undergo Systemic Therapy
Brief Title: Liver and Spleen Stiffness to Predict the Presence of Esaphageal Varices in Cirrhotic With Advanced HCC
Acronym: ELASTO-HCC
Status: Enrolling by invitation | Type: Observational
Sponsor: Azienda Ospedaliero Universitaria Policlinico Modena (Other)
Responsible Party: Principal Investigator, ANTONIO COLECCHIA, Prof of Gastroenterology, Azienda Ospedaliero Universitaria Policlinico Modena
Other Study IDs: AOU Policlinico Modena
Record Dates: First submitted 2025-01-09; First posted 2025-01-14 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-06

CONDITIONS: Hepatocellular Carcinoma; Liver Cirrhosis; Portal Hypertension
Keywords: HCC; Liver stiffness; Spleen stiffness; Esophageal varices; Portal Hypertension
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Cirrhosis; Hypertension, Portal; Esophageal and Gastric Varices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cirrhotic patients with advanced HCC: Cirrhotic patients with advanced HCC requiring systemic therapy will undergo upper endoscopy and measurement of liver and spleen stiffness.
  Interventions: Diagnostic Test: Liver and Spleen stiffness measurement.

INTERVENTIONS:
Diagnostic Test: Liver and Spleen stiffness measurement. — The use of spleen stiffness measurement to reduce unnecessary upper digestive endoscopies has never been evaluated in this patient setting.

SUMMARY:
Elasto-HCC is a prospective, uncontrolled, multicenter observational study involving several hepatology centers in Italy. Patients with liver cirrhosis and advanced hepatocellular carcinoma (HCC) who will need to undergo systemic therapy will be enrolled. Patients in the first phase will undergo measurement of liver and spleen stiffness and upper endoscopic evaluation and will subsequently be followed for 12 months

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) and clinically significant portal hypertension (CSPH) frequently coexist, affecting cirrhotic individuals' prognosis. Recently it has been confirmed that in cirrhotic patients with favorable Baveno VI consensus (platelets>150000/mm3 and liver stiffness measurement (LSM<20 kPa) or combined model based on spleen stiffness, endoscopic screening for varices could be avoided. The Portal Hypertension (PH)-related complications in all patients should be avoided and well managed, especially if they have advanced HCC (aHCC) at diagnosis. However, unlike patients without HCC, endoscopy is recommended for those who undergo systemic therapy, even if compatible with favorable Baveno VI consensus . The reasons for this indication derive from the consideration that the presence of HCC could influence the measurement of LSM and platelet count.

To date, in cirrhotic patients without HCC, according to Baveno VII consensus and the last EASL guidelines for non-invasive tests (NITs), besides LSM, Spleen Stiffness Measurement (SSM) is now considered the most accurate NITs for assessing portal hypertension and predicting the presence of esophageal varices (EVs) and varices needing treatment (VNT).

To date, no studies have evaluated the accuracy of NITs (LSM/SSM) on patients with advanced HCC (aHCC) who should undergo systemic therapy.

The study aims to assess the performance of SSM to rule out VNT in patients with aHCC who undergo systemic therapy.

Each center will prospectively collect data according to an electronic e-CFR on REDCap (Research Electronic Data Capture) system, a web application designed to support data capture for research studies in a secure manner.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 yrs;
* Cirrhotic patients of any etiology with aHCC scheduled to receive any line of systemic treatment for HCC;
* Patients are willing and able to give informed consent.

Exclusion criteria:

* Presence of splenic, mesenteric, or portal vein thrombosis.
* Previous placement of TIPS at the time of informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cirrhotic patients of any etiology with aHCC are scheduled to receive systemic treatment for HCC.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
: to evaluate the accuracy of Liver and Spleen stiffness in predicting the presence of high-risk EV needing treatment (VNT) in cirrhotic patients with aHCC who undergo systemic therapy. | from 2023 to 2025
  The patients at enrolment will be undergoing Upper endoscopy to assess the presence of esophageal or gastric varices and abdominal ultrasound (US) and contextual Liver and Spleen stiffness (LSM and SSM) with both Transient Elastography (FibroScan, Echosens) and a 2D-Shear-Wave Elastosonography to assess the Portal Hypertension (PH) degree; furthermore , biochemical analyses including platelet count (10^9/mm3), will also be performed

SECONDARY OUTCOMES:
Number of upper digestive endoscopies spared and Varices Needing Treatment (VNT) missed according to SSM/Baveno criteria evaluated | from 2023 to 2025
  According to Spleen stiffness measurement (SSM)/Baveno criteria, the number of upper endoscopies spared in patients without high-risk varices will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Pivetti, MD, Study Chair — Azienda Ospedaliera Universitaria Policlinico Modena; Luigi Colecchia, MD, Study Chair — IRCCS Azienda Ospedaliero-Universitaria, Bologna; Elton Dajti, MD, Study Chair — IRCCS Azienda Ospedaliero-Universitaria, Bologna
Locations (11):
- Italy (11):
  - UOC Gastroenterologia, Azienda Ospedaliero-Universitaria Policlinico Bari, Bari, Italy
  - UOC Gastroenterologia, IRCCS Policlinico Sant'Orsola, Università di Bologna, Bologna, Italy
  - UOC Medicina interna, malattie epatobiliari e immunoallergologiche, IRCCS Policlinico Sant'Orsola, Università di Bologna, Bologna, Italy
  - UOC Semeiotica Medica, IRCCS Policlinico Sant'Orsola, Università di Bologna, Bologna, Italy
  - Programma Dipartimentale di I fascia, Malattie del Fegato e delle vie Biliari, Azienda Ospedaliera Universitaria - Federico II, Università degli Studi di Napoli Federico II, Napoli, Napoli, Italy
  - Azienda Ospedaliera, Novara, Italy
  - UOC Clinica Medica 5 - Unit of Internal Medicine and Hepatology, Azienda Ospedale Università Padova,, Padua, Italy
  - UOC Centro Malattie Apparato Digerente (CEMAD, IRCCS Policlinico Agostino Gemelli, Università Cattolica del Sacro Cuore,, Roma, Italy
  - Dipartimento delle Scienze Mediche,Chirurgiche e Neuroscienze,UNISIEN, Siena, Italy
  - USD Liver Unit, Azienda Ospedaliera Universitaria Integrata Verona, Verona, Italy
  - UOC Gastroenterologia, Azienda Ospedaliera-Universitaria Policlinico di Modena, Modena

IPD SHARING:
Plan to Share IPD: Undecided